CLINICAL TRIAL: NCT03383562
Title: Daytime Variation of Complication in Gastric and Pancreatic Surgery : a Single Center Randomized Study
Brief Title: Daytime Variation of Complication in Gastric and Pancreatic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Chengfeng Wang, Director of Department of pancreatic and gastric Surgery, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: CT20180101
Record Dates: First submitted 2017-12-11; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Gastrointestinal Dysfunction; Hemorrhage; Infection; Fistula
MeSH Terms: conditions — Hemorrhage; Infections; Fistula | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- morning group: patients in the morning group are operated during 8:30 a.m. to 2:00 p.m.
  Interventions: Procedure: operation in different stages of the day
- afternoon group: patients in the morning group are operated during 2:00 p.m. to 8:00 p.m.
  Interventions: Procedure: operation in different stages of the day
- night group: patients in the morning group are operated during 8:00 p.m. to 12:00 p.m.
  Interventions: Procedure: operation in different stages of the day

INTERVENTIONS:
Procedure: operation in different stages of the day — operation was arranged in the morning ,afternoon or at night

SUMMARY:
Evaluate the daytime variation of complications in gastric and pancreatic surgery

DETAILED DESCRIPTION:
The trial is funded by Cancer Foundation of China. The trial is prepared to be registered on the clinicaltrails.gov. Quality assurance plan: every participant is enrolled or excluded by two practiced investigators. And two investigators participated in all steps of the trail, including the record of the data, and the investigators will compare the data. If the data is consistent, the investigators would record the data; if not, the data would be checked and decided by the two investigators. All the steps and data are site monitored and audited by the workers of research and financial department of National Cancer Center/ Cancer Hospital, Chinese Academy of Medical Sciences. Data check: the investigators compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry. Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources, including medical records and electronic case report forms. Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information, and normal ranges if relevant.

Standard Operating Procedures to address registry operations and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. All registry operations would be done according to specific steps, and by two practiced investigators. Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect. According to the formula to differ advantages and disadvantages, the investigators need at least 200 participants to take part in the trail.

The investigators can recruit about 600 participants every year according to previous experiences, so the investigators should recruit at least for half a year. Plan for missing data: the investigators would collect as much data as possible, and the investigators exclude the participants who cannot cooperate on recruitment. And the investigators manage situations according to statistical principles where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results. Statistical analysis plan: Kaplan-Meier method would be used to analyze the difference of complications between the three groups, and the local control rate of the three groups would be compared by chi square test. Statistical analyses would be performed by using International Business Machine Statistical Product and Service Solutions Statistics(version 20; IBM, Chicago, USA). The level of significance is defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo gastric or pancreatic surgery in our department.
2. Voluntary participation, Signing informed consent and have good compliance.

Exclusion Criteria:

1. Patient who attended other clinical trials in the last two months.
2. Patient who will undergo multiple organs resection.
3. Patient who has been taken anticoagulant recently.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who meet the inclusion criteria will be enrolled in this study and then will be arranged at morning ,afternoon or night group at random.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
gastrointestinal dysfunction | after operation from date of randomization until the date of first documented complications or date of death from any cause, whichever came first,up to 24 weeks
  using clinical symptoms to evaluate the gastrointestinal function after surgery
hemorrhage | after operation from date of randomization until the date of first documented complications or date of death from any cause, whichever came first, up to 24 weeks
  using clinical symptoms to evaluate the gastrointestinal function after surgery
infection | after operation from date of randomization until the date of first documented complications or date of death from any cause, whichever came first, up to 24 weeks
  using clinical symptoms to evaluate the gastrointestinal function after surgery
anastomotic fistula | after operation from date of randomization until the date of first documented complications or date of death from any cause, whichever came first,up to 24 weeks
  using clinical symptoms to evaluate the gastrointestinal function after surgery
test rating | after operation from date of randomization until the date of first documented complications or date of death from any cause, whichever came first, up to 24 weeks
  collecting blood sample to evaluate change of test after surgery

SECONDARY OUTCOMES:
Physical fitness index | after operation from date of randomization until the date of first documented complications or date of death from any cause, whichever came first,up to 24 weeks.
  The recovery of physical fitness index

CONTACTS AND LOCATIONS:
Overall Officials: Chengfeng Wang, B.A., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No